CLINICAL TRIAL: NCT03440515
Title: Management of Imatinib-associated Severe Skin Rash in Patients With Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1402
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Stromal Tumor(GIST)
Keywords: gastrointestinal stromal tumor; skin rash; imatinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Exanthema | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prednisone (Experimental): prednisone 30mg/day 3weeks oral, if on rash or pruritus prednisolone 20mg/day 3weeks -> 10mg/day->7.5mg/day->5mg/day->stop
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Prednisone treatment for severe skin rash induced by imatinib

SUMMARY:
To achieve optimal clinical outcomes with imatinib in GIST patients, it is crucial to maintain standard imatinib dose. Skin rash is a relatively common and sometimes severe adverse event of imatinib in GIST patients and may affect imatinib compliance. Our previous retrospective study suggested that severe skin rash induced by imatinib can be managed by systemic steroid without imatinib dose interruption or reduction. This phase II study was conducted to evaluate the efficacy and safety of systemic steroid in GIST patients with imatinib-associated severe skin rash.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older, at the time of acquisition of informed consent
* Histologically confirmed metastatic and/or advanced (unresectable or recurrent) GIST with CD117(+), DOG-1(+), or mutation in KIT or PDGFRα gene
* Patients with metastatic and/or advanced (unresectable or recurrent) GISTs, receiving imatinib as adjuvant or neo adjuvant, palliative chemotherapy for pre-or post- operations
* imatinib-associated severe skin rash which was defined as grade 3 skin rash or grade 2 skin rash with pruritus over grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
treatment success rate | 2 years
  Treatment success was defined as maintaining imatinib without persistence or recurrence of skin rash requiring 1) additional systemic steroid treatment, and 2) interruption or dose reduction of imatinib.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim EJ, Ryu MH, Park SR, Beck MY, Lee WJ, Lee MW, Kang YK. Systemic Steroid Treatment for Imatinib-Associated Severe Skin Rash in Patients with Gastrointestinal Stromal Tumor: A Phase II Study. Oncologist. 2020 Nov;25(11):e1785-e1793. doi: 10.1634/theoncologist.2019-0953. Epub 2020 Jul 12. PMID 32589310